CLINICAL TRIAL: NCT02125175
Title: BIOPROP20: Biologically Optimised IMRT for Prostate Radiotherapy Hypofractionated Radiotherapy With Intra-prostatic Boosts to Tumour Nodules in Men With Intermediate and High Risk Prostate Cancer
Acronym: BIOPROP20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDD547
Record Dates: First submitted 2014-04-17; First posted 2014-04-29 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hypofractionated IMRT boost Radiotherapy (Experimental)
  Interventions: Radiation: Hypofractionated IMRT boost Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated IMRT boost Radiotherapy

SUMMARY:
High dose radiotherapy is a very effective treatment for prostate cancer. However, there is an increased risk of side effects compared to lower dose radiotherapy. This study will investigate the use of dose painting radiotherapy. Dose painting radiotherapy administers a high dose of radiotherapy to areas of cancer inside the prostate and a lower (standard) dose to the rest of the prostate. This may improve control of the cancer without increasing the side effects. The radiotherapy is given in 20 doses, called fractions.

DETAILED DESCRIPTION:
For patients with prostate cancer which has not spread, the typical treatment is hormone therapy and radiotherapy.

It is possible to identify areas within the prostate which contain a significant amount of cancer with functional MRI or with 18F choline PET CT scans. These areas are called Dominant Intraprostastic Lesions 'DILs'. Targeted prostate biopsies help to confirm scan results. The radiotherapy dose to the DILs is increased, whilst the rest of the prostate is treated with the standard dose. This technique is called dose painting or 'boost' Intensity Modulated Radiotherapy Treatment (IMRT).

IMRT is given in 37 treatment doses called fractions, once a day for about 8 weeks. A hypofractionated schedule is the administration of the total radiotherapy treatment over a smaller number of fractions, at a higher dose per fraction. Recent evidence suggests that the idea of using a 'hypofractionated' treatment schedule is better and more convenient with a similar number of side effects as a regular schedule.

In the study, 50 patients with intermediate/high risk prostate cancer suitable and fit for radical radiotherapy will be recruited. The patients undergo a staging functional MRI scan, fiducial marker insertion (required for image guided radiotherapy) and hormone therapy as per standard of care treatment. The choline PET CT scan and targeted prostate biopsies are optional. They are useful if the MRI is difficult to interpret and will be offered to patients if they are felt to be appropriate by the clinician. After 2 months hormone therapy (standard protocol) patients have a CT /MRI planning scan and undergo IMRT with 20 treatments (fractions).The patient will then be followed up until 24 months after they started radiotherapy treatment.

The main aim is to assess the side effects related to the bladder and bowel at 18 weeks (acute toxicity) after starting hypofractionated IMRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate
2. NCCN intermediate/high risk disease and estimated risk of lymph node involvement 15 - 40%*
3. MRI stage T2a-T4 N0M0
4. Age 18-80 years
5. Normal blood count (Hb >11g/dl, WBC > 4000/mm3, platelets >100,000/mm3)
6. WHO performance status 0 or 1
7. Fully informed written consent

   * Risk of pelvic lymph node involvement = (Gleason score - 6) x 10 + 2/3 PSA

Exclusion Criteria:

1. Prior radiotherapy to the prostate or pelvis
2. Prior hormone therapy or radical prostatectomy
3. Total hip replacement
4. Clinically significant inflammatory bowel disease
5. Contraindication to have diagnostic MRI scans
6. Unable to have a general anaesthetic
7. Anti-coagulant therapy which cannot be temporarily stopped

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-01; Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Acute bladder and bowel toxicity (NCI CTCAE v 4.0 and RTOG) at 18 weeks after the commencement of radiotherapy treatment | 18 weeks

SECONDARY OUTCOMES:
The success rate of producing dose painted IMRT plans which fulfill the dose-volume constraints as specified for the prostate and for the normal tissues | 3 years
Late bladder and bowel toxicity (NCI CTCAE v4) at 2 years | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Syndikus, MD, Principal Investigator — The Clatterbridge Cancer Centre NHS Foundation Trust
Locations (1):
- The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral, United Kingdom

REFERENCES:
- [Derived] Chatterjee R, Chan J, Mayles H, Cicconi S, Syndikus I. Long-term Results of Hypofractionated Radiotherapy With Intra-prostatic Boosts in Men With Intermediate- and High-risk Prostate Cancer: A Phase II Trial. Clin Oncol (R Coll Radiol). 2024 Dec;36(12):e473-e482. doi: 10.1016/j.clon.2024.08.011. Epub 2024 Aug 22. PMID 39242247
- [Derived] Onjukka E, Uzan J, Baker C, Howard L, Nahum A, Syndikus I. Twenty Fraction Prostate Radiotherapy with Intra-prostatic Boost: Results of a Pilot Study. Clin Oncol (R Coll Radiol). 2017 Jan;29(1):6-14. doi: 10.1016/j.clon.2016.09.009. Epub 2016 Sep 29. PMID 27692920